CLINICAL TRIAL: NCT03806153
Title: Do the Morphokinetic Parameters of Early Embryonic Development Have an Interest in the Choice of the Embryo to be Transferred and Improve Birth Rates in Vitro Fertilization
Brief Title: Interest of Morphokinetic Parameters of Early Embryonic Development in the Birth Rates in Vitro Fertilization
Acronym: EMCIMO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017/385/HP
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Reproductive Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional morphology arm (reference method) (Active Comparator)
  Interventions: Other: Morphokinetic
- Morphokinetic arm (Experimental)
  Interventions: Other: Morphokinetic

INTERVENTIONS:
Other: Morphokinetic — The embryos will be observed at a fixed time and according to morphological criteria (Alpha Specialist Group in Reproductive Medicine and ESHRE, 2011). and all the films obtained will be analyzed. Embryos will be classified according to morphokinetic criteria (Ciray et al., 2014).

SUMMARY:
In France, nearly 3% of children are conceived by the technique of Assisted Reproductive Medicine, of which nearly 70% by in vitro fertilization (IVF). The rates of clinical pregnancy by oocyte retrieval or embryo transfer have not changed much. The use of mono-embryo transfer reduces the risk of multiple pregnancies and associated obstetric complications. The choice of embryo to transfer or freeze is a key element in improving the chances of success of IVF. It is usually based on conventional morphological criteria (reference method) that are punctual, qualitative and subjective. However, embryo morphology at early stages has little predictive value for obtaining a late-stage embryo and its chances of implantation. The recent use of time-lapse technology during embryonic culture makes it possible to associate morphological criteria with continuous monitoring of the kinetics of embryonic development. The choice of the embryo to be transferred is then made according to morphokinetic criteria (conventional morphological criteria to which are added the data of the kinetics of embryonic development).

Two recent retrospective studies give contradictory results, the first shows higher birth rates in the group of embryos selected according to conventional morphological criteria, the second concludes that morphokinetic analysis is superior. Morphokinetic criteria would also be more objective and reproducible. However, the use of morphokinetic parameters remains controversial in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. For the couple:

   * Couple whose two members are 18 years old and over,
   * Couple whose two members are affiliated to a social security scheme,
   * Couple whose two members read and understood the newsletter and signed the consent form for their participation in this research.
2. For the conditions of realization of the ICSI attempt:

   * Couple supported for a 1st or 2nd attempt at in vitro fertilization with sperm microinjection (ICSI) for male infertility,
   * In vitro fertilization attempt performed with micro-injection of fresh ejaculated spermatozoa.
3. For the man:

   * Couple whose man has an alteration of at least one of the sperm parameters according to the WHO (WHO, 2010) for the number, concentration, vitality, mobility or morphology according to the modified David classification (Auger and Eustache, 2000).

Exclusion Criteria:

1. For the couple:

   * Couple whose wife is under 18 and over 42 and / or the male is under 18 and over 59
   * Couple already included in the protocol "EMCIMO" for a previous attempt,
   * Couple of which one or both members is deprived by an administrative or judicial decision or subject to a legal measure of protection of the majors (safeguard of justice or tutelage or curatorship),
   * Couple where one or both members do not speak or understand French.
2. For the conditions of realization of the ICSI attempt:

   - In vitro fertilization attempt with the micro-injection of testicular spermatozoa, epididymal, previously frozen or resulting from a retrograde ejaculation.
3. For the man:

   * Severe oligozoospermia (<100,000 spermatozoa / ejaculate).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 520 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study will be the live birth rate by fresh embryo transfer(s). | 36 months